CLINICAL TRIAL: NCT02827149
Title: High Resolution Donor Recipient HLA Matching Level in Unrelated Hematopoietic Stem Cell Transplantation and Impact on the Transplant Outcome: the Italian Experience
Brief Title: High Resolution Donor Recipient HLA Matching Level in Unrelated HSCT
Acronym: GITMO-HLA-HR
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Trapianto di Midollo Osseo (Other)
Collaborators: Associazione Italiana di Immunogenetica e Biologia dei Trapianti (AIBT) (Unknown); National Marrow Donor Program (Other); University of Rome Tor Vergata (Other)
Responsible Party: Sponsor
Other Study IDs: GITMO-HLA-HR
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Hematologic Diseases
Keywords: HSCT; high resolution HLA typing; unrelated donor
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Italian, retrospective, prospective, observational, multicentre, spontaneous, non-interventional, non-pharmacological The study aims to analyze in the national Italian experience

1. The compatibility level selected by the Italian Transplant Centres using an high resolution HLA typing at the start of search process for hematopoietic stem cell transplantation from volunteer unrelated donor
2. The transplant outcomes in terms of Overall Survival, Disease Free Survival, Relapse Rate and Transplant Related Mortality and the correlation with the level of HLA matching pairs of donor/recipient included in the Italian Bone Marrow Donor Registry and Promise registry.
3. The possible identification of allelic mismatching combinations characterized by increased cross-reactivity associated with higher incidence of acute or chronic graft-versus-host disease .
4. The possible identification of combinations of allelic mismatching characterized by higher permissiveness.

DETAILED DESCRIPTION:
Haematopoietic allogeneic stem cell transplantation (HSCT) represents a potentially curative treatment for several haematological disorders, but its application depends on the availability of a suitable donor. Some data show that in US population the likelihood of finding HR 8/8 HLA A, B, C, DRB1 matched donor in NMDP registry is about 75% for white Europeans but only 46% for white patients of Middle Eastern or North African descents. Moreover, this probability decreases for patients belonging to African or Black South/Central American group at 18% and 16%, respectively. Furtherly, recent data have reported a significant improvement in the unrelated donor identification over the years. In particular, they have conducted the unrelated donor searches for 1344 ideal patients in the "Be The Match Registry" database at 2 time points: 2009 and 2012. Their results have shown that 8/8 high resolution HLA match rate (A, B, Cw and DRB1) for White raised from 68% in 2009 to 72% in 2012. Corresponding match rates were 41% to 44% for Hispanic, 44% to 46% for Asian/Pacific Islander), and 27% to 30% for African American/Black race and ethnic groups for 2009 and 2012, respectively. The 2012 10/10 match rates were 67% for White, 38% for Hispanic, 41% for Asian/Pacific Islander, and 23% for African American/Black.

Current available data confer to HLA mismatch (6-7/8) a significant increased risk for grades II to IV and III to IV acute graft versus host disease, chronic graft versus host disease, transplant-related mortality (TRM) and overall mortality compared with HLA-matched cases (8/8). However, it is not yet clear if type (allele/antigen) and locus (HLA-A, -B, -C, and -DRB1) of mismatch are associated with overall mortality. In order to improve the outcome of the unrelated HSCT, many efforts are ongoing for identifying permissive and non permissive HLA disparity both for I and II classes HLA. Recently, several authors have highlighted the crucial role of allelic mismatching Cw combinations in supporting GVL/ graft versus host disease effect with a consequent decreased risk of relapse (p<0.003). On the contrary, Cw disparities as Cw03:03 vs Cw03:04 or Cw07:01 vs Cw07:02 seem to be permissiveness in terms of HSCT clinical outcome. Contemporarily, Japanese meta-analysis on 6967 unrelated HSCT has shown that the presence of HLA-B*51:01 in the donor/recipient pairs is associated with acute graft versus host disease not only for the strong linkage disequilibrium of HLA-C*14:02 and -B*51:01 but also for the effect of HLA-B*51:01 itself. Based on these data, mismatched HLA-C*14:02 should be considered a non-permissive HLA-C mismatch in donor selection because it seems to be a potent risk factor for severe acute graft versus host disease and mortality.

Concerning DPB1 HLA loci, an algorithm for non-permissive HLA-DPB1 disparities has been described, based on T-cell alloreactivity patients, with potential clinical implications. To confirm this data, GITMO analysis has reported an increased but similar overall mortality by non-permissive HLADPB1 disparity in 10 of 10 (HR 2.12; CI, 1.23-3.64; P .006) and 9 of 10 allele-matched transplantations (HR 2.21; CI, 1.28-3.80; P .004), both in early-stage and in advanced-stage disease. Additionally, recent data have reported that among 8/8 matched cases, HLA-DPB1 and -DQB1 mismatch resulted in increased acute graft versus host disease and HLA-DPB1 mismatch is associated with decreased relapse. Non-permissive HLA-DPB1 allele mismatch was also associated with higher TRM compared with permissive HLA-DPB1 mismatch or HLA-DPB1 match and increased overall mortality compared with permissive HLA-DPB1 mismatch in 8/8 (and 10/10) matched cases. Based on all these reports, the current suggestions concerning the unrelated donor selection consists of a full matching at HLA-A, -B, -C, and -DRB1 unrelated donor for optimal HSCT survival, and avoiding non-permissive HLA-DPB1 mismatches in otherwise HLA-matched pairs.

In 2009, a previous retrospective Italian analysis, performed on 805 couples, reported that globally there are no differences in terms of outcomes (Overall Survival, Disease Free Survival, Relapse Rate and Transplant Related Mortality and Graft Versus Host Disease) in adult patients with neoplastic diseases transplanted with HLA-matched donor 10/10 or 9/10. However, stratifying patients by stage of disease at transplant, a single HLA incompatibility significantly increases the risk of mortality in patients who received HSCT in early stage whereas this data is not confirmed for patients transplanted in advanced stage of disease. This previous Italian analysis included only 10/10 high-resolution typed pairs from 1999 to 2006, excluding all the others couple without a full HLA typing for avoiding confounding results. According to Italian Bone Marrow Donor Registry standard, extended HR HLA was not a mandatory requirement from 1999 to 2006.

From January 2012, all Italian recipients have been typed with HR-HLA typing at the starting of the unrelated donor search process with a consequent advantage in terms of "non selected population" as object of the present observational trial. Moreover, the larger size of cohort of patients who underwent unrelated HSCT during a smaller study period of 2 years should lead to a more effective analysis including the assessments of permissive and non-permissive I and II class HLA incompatibilities. Finally, in order to give a stronger statistical power to this trial, particular efforts have been drawn in order to recovery data about the graft versus host disease prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

Haematological disease

Written and signed PROMISE informed consent

Patient undergoing unrelated HSCT

Exclusion Criteria:

Unavailability of HR-HLA pairs typing including at least A, B, C, DRB1 loci

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enrol adult patients who received hematopoietic stem cell transplantation (HSCT) from unrelated adult donor between 1° January 2012 and 31 December 2015.
Sampling Method: Probability Sample
Enrollment: 1838 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-21 (Actual)

PRIMARY OUTCOMES:
compatibility level | 4 months by Activation of the donor search
  The compatibility level selected by the Italian Transplant Centres using an high resolution HLA typing at the start of search process for Hematopoietic Stem Cell Transplantation from volunteer unrelated donor
Overall survival from transplant | 100 days, 1 year and 2 years from transplant
  The transplant outcomes in terms of Overall Survival and the correlation with the level of HLA matching pairs of donor/recipient included in the Italian Bone Marrow Donor and Promise Registry.
Disease Free Survival | 100 days, 1 year and 2 years from transplant
  The transplant outcomes in terms of Disease Free Survival and the correlation with the level of HLA matching pairs of donor/recipient included in the Italian Bone Marrow Donor and Promise Registry
Relapse Rate | 100 days, 1 year and 2 years from transplant
  The transplant outcomes in terms of Relapse Rate and the correlation with the level of HLA matching pairs of donor/recipient included in the Italian Bone Marrow Donor and Promise Registry.
Transplant Related Mortality | 100 days, 1 year and 2 years from transplant
  The transplant outcomes in terms of Transplant Related Mortality and the correlation with the level of HLA matching pairs of donor/recipient included in the Italian Bone Marrow Donor and Promise Registry.

SECONDARY OUTCOMES:
identification of allelic mismatching | 2 years from transplant
  The possible identification of allelic mismatching combinations characterized by increased cross-reactivity associated with higher incidence of acute or chronic GVHD.
identification of allelic mismatching | 2 years from transplant
  2. The possible identification of combinations of allelic mismatching characterized by higher permissiveness.
Acute Graft-versus-Host Disease (aGvHD) | from date of transplant to until the date of first event of aCGVD assessed up to 100 days post transplant]
  The available information in the EBMT data regard the date of onset and the maximum grade of aGvHD. It is therefore possible to estimate the probability of aGvHD in a competing risks setting (death is a competing event; whether relapse/progression is a competing event must be discussed with the physician). By definition, patients alive (relapse/progression-free) at day 100 without having experienced aGvHD are censored. If the dates of onset are missing for the majority of patients, the analysis can focus only on the occurrence of aGvHD, which is analyzed by a logistic regression model. This method would however be incorrect if there is a (non negligible) percentage of censored observations or if competing events occurred before day 100.
Chronic Graft-versus-Host Disease (cGvHD) | from day +100 post transplant to until the date of first event to cGVHD assessed up to 2 years post enrolment]
  When possible, if information on the date of 1°occurrence of cGvHD is available, it should be analyzed as a time-to-event outcome, being death (and possibly relapse/progression) the competing event; data are censored for patients alive (relapse/progression-free) without episodes of cGvHD at last follow-up. Since cGvHD is defined only for patients surviving at least 100 days, the survival model should consider a left truncation at 100 days; alternatively, the time of occurrence of cGvHD must be computed from 100 days. If information on the timing of cGvHD is not available, the outcome considered is the occurrence, and the statistical model to be used is the logistic regression. Only patients surviving at least 100 days are considered to be at risk of developing cGvHD, therefore the analysis must be restricted to these patients. This analysis is of course not satisfactory because it does not take into account the occurrence of death and censoring.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Picardi, MD, Principal Investigator — Policlinico Università Tor Vergata - Rome
Locations (39):
- Italy (39):
  - Azienda Ospedaliera SS Antonio e Biagio, Alessandria
  - Clinica di Ematologia - Ospedali Riuniti di Ancona, Ancona
  - Ospedale Mazzoni, Ascoli Piceno
  - Policlinico di Bari-Ematologia con trapianti, Bari
  - Divisione di Ematologia - Ospedali Papa Giovanni XXIII, Bergamo
  - Ospedale San Orsola, Bologna
  - AO Spedali Civili di Brescia- USD - TMO Adulti, Brescia
  - Ospedale Binaghi, Cagliari
  - Ospedale Ferrarotto - Ematologia, Catania
  - S.C. Ematologia - Azienda Ospedaliera S. Croce e Carle, Cuneo
  - Cattedra di Ematologia - Azienda Ospedaliera di Careggi, Florence
  - Ematologia e Centro Trapianti Midollo Osseo - Ospedale IRCCS Casa Sollievo della Sofferenza, Foggia
  - AOU IRCCS San Martino - IST, Genova
  - Divisione di Ematologia - Istituto Nazionale dei Tumori, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - IEO, Milan
  - Ospedale San Raffaele, Milan
  - Divisione Ematologia - Azienda Ospedaliera Universitaria - Policlinico -, Modena
  - Ospedale San Gerardo, Monza
  - A.O.U. Policlinico Federico II, Napoli
  - AO Ospedali Riuniti Villa Sofia - Cervello, Palermo
  - Dipartimento Oncologico La Maddalena, Palermo
  - Fondazione IRCCS San Matteo, Pavia
  - Policlinico San Matteo, Pavia
  - Dip. Medicina Clinica e Sperimentale, Perugia
  - Ospedale Civile, Pescara
  - Ospedale G. Da Saliceto di Piacenza, Piacenza
  - Centro Unico Regionale Trapianti di Midollo Osseo - Ospedale Bianchi-Melacino-Morelli, Reggio Calabria
  - A.O. San Camillo Forlanini, Roma
  - Cattedra di Ematologia - Policlinico, Roma
  - Divisione di Ematologia - Istituto di Semeiotica Medica - Policlinico A. Gemelli, Roma
  - Policlinico Universitario Tor Vergata, Roma
  - Dipartimento di Oncologia Medica ed Ematologia - Istituto Clinico Humanitas, Rozzano (MI)
  - Ospedale Moscati, Taranto
  - AOU CIttà della Salute e della Scienza, Torino
  - Ospedale Regina Margherita, Torino
  - Clinica Ematologica - AOU Santa Maria Della Misericordia, Udine
  - AOU Integrat, Verona
  - Ospedale S. Bortolo-Divisione Ematologia, Vicenza